CLINICAL TRIAL: NCT01964885
Title: Clinical Trial to Explore Benefit and Tolerability of IQP-AS-105 (Xaludicin®) in Subjects With Increased Susceptibility to Upper Respiratory Tract Infections
Brief Title: Benefit and Tolerability of IQP-AS-105 in Reducing Susceptibility to Upper Respiratory Tract Infections
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: No significant results during interim analysis
Sponsor: InQpharm Group (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: INQ/012213
Record Dates: First submitted 2013-10-15; First posted 2013-10-17 (Estimated); Last update posted 2016-02-12 (Estimated); Status verified 2016-02

CONDITIONS: Common Cold; Upper Respiratory Tract Infections
MeSH Terms: conditions — Common Cold; Respiratory Tract Infections

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- IQP-AS-105 (Active Comparator): One tablet daily
  Interventions: Dietary Supplement: IQP-AS-105
- Placebo (Placebo Comparator): One tablet daily
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: IQP-AS-105
  Arms: IQP-AS-105
Dietary Supplement: Placebo
  Arms: Placebo

SUMMARY:
IQP-AS-105, is a food supplement derived from garlic (Allium sativum). The objective of this study is to evaluate the possibilities of clinical use of IQP-AS-105 as a preventive medicine, based on its ability to enhance the immune system responses

ELIGIBILITY:
Inclusion Criteria:

* age 18-70 years
* increased risk for infections - at least 4 cold episodes within 12 months
* commitment to adhere to their accustomed diet and physical activity
* women of child-bearing potential have to agree to use appropriate birth control methods
* written consent of the subject to participate is a prerequisite for study participation

Exclusion Criteria:

* acute / chronic upper airways disease
* chronic cough of any origin
* acute / chronic lower airways disease
* any allergic reaction that may influence the study outcome (e.g. acute/chronic rhinitis)
* history of nasal reconstructive surgery
* presence of nasal ulcers or nasal polyps
* severe nasal septum deviation or other condition that could cause nasal obstruction
* congenital or acquired immunodeficiency disease (e.g. HIV infection)
* severe organ or systemic diseases
* body temperature above 37.5°C
* suspected swine flu or influenza
* vaccination against influenza or swine flu within 3 months prior to study start
* stomach/gastrointestinal diseases
* sleep disorder
* psychiatric disorders
* known sensitivity to the ingredients of the investigational product
* intake of products that may influence the study outcome within the last 14 days prior to study start and during the study
* analgesics , antibiotics or decongestant nose drops/spray, unless they are used as rescue medications
* pregnancy or nursing
* alcohol / drug abuse
* simultaneous participation in another clinical trial or participation in a clinical trial within the last 30 days
* insufficient compliance

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2013-10; Primary Completion 2014-04 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Difference in severity of common cold symptoms for cold episodes between the two arms | 12 weeks
  Assessed by WURSS-21

SECONDARY OUTCOMES:
Incidence of cold episodes | 12 weeks
Duration of cold episodes | 12 weeks
Severity of cold symptoms over the first 4 days of the episode | 12 weeks
Severity of cold symptoms over the first 7 days of the episode | 12 weeks
Day and score value of the maximal WURSS-21 daily score | 12 weeks
Severity of cold somptoms from the date of the maximal WURSS-21 daily score, for 4 days following thereafter | 12 weeks
Incidence of viral infection | 12 weeks
Use of rescue medication | 12 weeks
Number of days on sick leave related to cold episodes | 12 weeks
Number of re-infections | 12 weeks
Severity of cold symptoms at first episode | 12 weeks
Severity of cold symptoms at recurring (subsequent) episodes | 12 weeks
Severity of cold episodes during the 4 week follow-up period | 12 weeks
Changes in special laboratory parameters in the subgroup | 7 days
Changes in cytokine production in the subgroup | 7 days
global evaluation of the benefit by the subjects / investigators | 12 weeks
Global assessment of tolerability by subjects/investigators | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Udo Bongartz, PhD, Principal Investigator
Locations (1):
- Udo Bongartz, Berlin, State of Berlin, Germany